CLINICAL TRIAL: NCT05941676
Title: Evaluation of the Prognostic Potential of New Immune Biomarkers in Non-metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Prognostic Immune Biomarkers in HNSCC
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: ONKOL-01-Head and neck; RVO-FNOs/2021 (Other Grant/Funding Number: University Hospital Ostrava)
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma
Keywords: immune biomarkers; tumor-infiltrating lymphocytes; PD-L1 (programmed death ligand-1) expression; prognosis; head and neck cancer; head and neck squamous cell carcinoma (HNSCC); radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy specimen from the primary tumour in head and neck, before curative radiotherapy/radiochemotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck carcinoma patients: Head and neck carcinoma patients will be enrolled in this study group.
  Interventions: Diagnostic Test: Tumour immunoprofile evaluation

INTERVENTIONS:
Diagnostic Test: Tumour immunoprofile evaluation — Tumour immunoprofile evaluation will be performed in patients with head and neck cancer.

SUMMARY:
Evaluation of the prognostic potential of tumor-infiltrating lymphocytes and PD-L1 expression in non-metastatic squamous cell carcinoma of the head and neck

DETAILED DESCRIPTION:
The role of the immune system in the process of tumor growth and progression in head and neck (HaN) cancer has become of increasing importance. In the last years, the concept of tumor immune microenvironment (TIME) with the presence of tumor cells (TC) and infiltrating immune cells (IC) has been intensively studied. The results of available clinical studies suggest a positive impact of tumor-infiltrating lymphocytes (TILs) on the prognosis of HNSCC patients and their overall (OS) and cancer specific survivals. Beside TILs, an integral component of TIME is the immunosuppressive activity represented by inhibitory signalling molecules expressed on tumor cells (TCs) and immune cells (ICs).

One of these molecules is programmed death-ligand 1 (PD-L1), which inhibits the cytotoxic immune response mediated by T-lymphocytes.

The aim of this observational cohort study is to assess the prognostic potential of novel immune biomarkers in patients with HNSCC tumors stage I-IVb treated with radical radiotherapy and radiochemotherapy. Specifically, the association between high and low TILs infiltration and OS and cancer specific survival parameters will be investigated. As well as the association between high and low PD-L1 expression and OS and cancer specific survival parameters will be investigated.

This is a non-interventional study conducted in one institution - Department of oncology, University hospital Ostrava. The tumor immunoprofile defined by the presence of immune biomarkers (TIL, PD-L1) will be evaluated in each patient from biopsy specimens in representative hematoxylin and eosin stained sections by immuno-histochemistry. The Cox proportional risk model will be used to estimate the prognostic potential of each of the biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-metastatic squamous-cell head and neck cancer (HNSCC) stage I-IVb indicated for curative/radical treatment
* Histologically verified squamous cell carcinoma including HPV-positive carcinomas
* Tumor site: oropharynx, larynx, hypopharynx, oral cavity, nasal cavity
* Treatment modality - radiotherapy or radiochemotherapy
* Presence of immune biomarkers in the tissue - tumor-infiltrating lymphocytes (TILs) and/or PD-L1 expression
* Sufficient data on patient follow-up

Exclusion Criteria:

* Histological type other than squamous cell carcinoma
* Paranasal sinus tumors, thyroid and nasopharyngeal carcinomas, salivary gland tumors, mucosal melanoma, skin carcinoma, lymphomas, and occult primary tumors
* Synchronous malignancies or recurrent disease
* The previous use of radiotherapy
* The presence of distant metastatic disease
* Missing or inadequate follow-up data
* The inability to evaluate biomarkers (TILs or PD-L1) in a histological tissue sample.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stage I-IVb HNSCC indicated for radical treatment - radiotherapy or radiochemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 24 months
  Overall survival measured in months - calculated from the date of initiation of radiotherapy to the date of death from any cause or the date of the last follow-up visit.

SECONDARY OUTCOMES:
Disease-specific survival (DSS) | 24 months
  Disease-specific survival calculated from the date of initiation of radiotherapy to the date of cancer death, or date of the last follow-up visit. Patients who died from causes other than HNSCC are censored at the time of death.
Disease-free survival (DFS) | 24 months
  Disease-free survival calculated from the date of initiation of radiotherapy to the date of detection of any recurrence, or date of death from any cause or date of the last follow-up visit. Patients without tumor recurrence are censored at the last follow-up contact.
Locoregional-free survival (LRFS) | 24 months
  Locoregional-free survival calculated from the date of initiation of radiotherapy to the date of detection of clinical, radiological and/or pathological evidence of recurrence or tumor progression at the primary site or in the regional nodal area, or date of death from any cause or date of the last follow-up visit. Patients without tumor recurrence are censored at the last follow-up contact.
Distant metastatic-free survival (DMFS) | 24 months
  Distant metastatic-free survival calculated from the date of initiation of radiotherapy to the date of detection of distant metastasis of the tumor, or date of death from any cause or date of the last follow-up visit. Patients without tumor recurrence were censored at the last follow-up contact.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Result] Blazek T, Petras M, Knybel L, Cvek J, Soumarova R. Programmed Cell Death Ligand 1 Expression on Immune Cells and Survival in Patients With Nonmetastatic Head and Neck Cancer: A Systematic Review and Meta-analysis. JAMA Netw Open. 2023 Mar 1;6(3):e236324. doi: 10.1001/jamanetworkopen.2023.6324. PMID 37000447
- [Derived] Blazek T, Petras M, Hurnik P, Matousek P, Knybel L, Cermakova ZZ, Stembirek J, Cvek J, Soumarova R. High PD-L1 expression on immune cells along with increased density of tumor-infiltrating lymphocytes predicts a favorable survival outcome for patients with loco-regionally advanced head and neck cancer: early results from a prospective study. Front Oncol. 2024 Apr 4;14:1346793. doi: 10.3389/fonc.2024.1346793. eCollection 2024. PMID 38638854